CLINICAL TRIAL: NCT01326572
Title: Prevalence and Pathogenesis of Lung Disease in a Large HIV Cohort-Pitt
Brief Title: Lung HIV Disease in a Large Cohort-Pitt
Acronym: MACS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of California, Los Angeles (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: LUNG007; 5R01HL090339 (NIH)
Record Dates: First submitted 2011-02-21; First posted 2011-03-31 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2016-05

CONDITIONS: Pulmonary Disease; HIV; Emphysema
Keywords: HIV; Pulmonary disease; emphysema; COPD
MeSH Terms: conditions — Lung Diseases; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, sputum, oral wash, bronchial washes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- female, male, HIV, lung disease: All participants in the University of Pittsburgh Multicenter AIDS Cohort Study are eligible for this protocol. All participants in the UCSF Women's HIV study are eligible and all Men from the UCLA men's HIV study are eligible

SUMMARY:
HIV-infected patients have an increased incidence of emphysema compared to non-HIV-infected patients, and it has been hypothesized that this accelerated disease progression is the result of one or more latent infections that amplifies the pulmonary inflammatory response. The investigators will examine the prevalence and progression of emphysema in subjects with and without HIV and determine risk factors for emphysema in this population.

DETAILED DESCRIPTION:
Specific Aim 1: To test the hypothesis that emphysema is more prevalent and progresses more quickly in HIV+ subjects compared to HIV- controls: The investigators will characterize the prevalence, nature, and progression of HIV-associated emphysema. Emphysema will be determined in HIV+ and HIV- subjects by spirometry, diffusing capacity, and quantitative computed tomography and/or EBCT. These studies will be repeated at 18 and 36 months after baseline to assess differences in progression between HIV+ and HIV- subjects. Multifactorial regression analyses will determine the contribution of various risk factors to presence and progression of emphysema.

The investigators will perform pulmonary function testing at baseline and compare degree of obstruction according to HIV status while adjusting for other clinical variables that influence lung function. Assessment of degree of emphysema and its distribution can be accomplished using quantitative CT morphometry density analysis. This technique measures lung density by pixel analysis expressed in Hounsfield units (HU) or its inverse (ml of gas/gram of tissue) which increases proportionately with the magnitude of emphysema. These measurements have been histologically-verified and give quantitative, reproducible measurements of percentage and distribution of lung considered normal, mildly emphysematous, and severely emphysematous. The investigators will compare emphysema in the HIV+ and HIV- subjects and compare progression over time.

Specific Aim 2: To establish a bank of saliva, sputum, serum, plasma, DNA, RNA, proteins and cells from the biological samples of these subjects with a purpose of performing future proteomic and genomic analyses of gene expression, genetic associations, disease pathogenesis and markers of disease progression in subjects with HIV infection and lung diseases:

2a) To test the role of low level infections with physiologic obstruction in HIV-infected patients. The investigators will examine the role of co-infection with Pneumocystis and other microbes in the pathogenesis of HIV-associated emphysema and the mechanism by which they cause emphysema progression by examining induced sputum specimens at baseline, 18 months, and 36 months.

Specific Aim 3. To test the hypothesis that persistent, sub-clinical infection in HIV+ subjects augments the pulmonary inflammatory response and leads to emphysema.

3a. To test the hypothesis that pulmonary colonization is increased in subjects with HIV-associated emphysema. The investigators will perform serial bronchoscopic alveolar lavage (BAL) in four groups of HIV+ and HIV - subjects: smokers with emphysema, smokers without emphysema, non-smokers with emphysema, and non-smokers without emphysema at the four sub-study sites. The investigators will use culture and molecular techniques to test for pathogens associated with emphysema and/or HIV and compare results between groups at baseline and over time to test our hypothesis that HIV+ subjects with emphysema harbor sub-clinical infection and that these infections accelerate lung damage and inflammation. The investigators will also determine pulmonary HIV levels and their relationship to emphysema and colonization.

3b. To test the hypothesis that local inflammatory responses and proteases are upregulated in HIV+ subjects with emphysema. BAL cellular infiltration will be characterized by flow cytometry to develop a quantitative and qualitative evaluation of cellular inflammatory responses in the four patient groups in Aim 3a. Lymphocyte populations will be analyzed for activation markers and intra-cellular cytokine production. The investigators will measure cytokine expression and protease levels in BAL supernatant as well as macrophage protease production. The investigators will compare results between groups and correlate with infections and HIV BAL viral levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* By participant's report, s/he is:
* HIV positive OR
* HIV negative and at high risk
* Recruited via:
* Pitt Men's Study/MAC
* Women's Interagency Health Study
* Attendee of UPMC HIV/AIDS Program

Exclusion Criteria:

* Acute onset of shortness of breath, cough, fever or heart condition such as tachycardia, angina or arrhythmias
* Pregnancy
* MI, CVA or cardiovascular event within last 3 months
* Eye or abdominal surgery with last 3 months
* Active TB by documentation or self-report
* Weight > 500 lbs.
* Exposure to > 10 rads in the previous 12 months (i.e., 2 CT or 4 cardiac cath…or other fluoroscopic exams For bronchoscopy subjects only
* Subjects with an upper or lower respiratory tract infection
* Individuals with a Primary diagnosis of vocal cord dysfunction, or those with significant or uncontrolled systemic diseases will be excluded
* 75 years of age or older

Ages: 18 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinic for Pittsburghs Mens Aids Clinic Study(MACS)
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2009-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The investigators will compare emphysema in the HIV+ and HIV- subjects and compare progression over time. | 36 months
  The investigators will perform pulmonary function testing at baseline and compare degree of obstruction according to HIV status while adjusting for other clinical variables that influence lung function. Assessment of degree of emphysema and its distribution can be accomplished using quantitative CT morphometry density analysis. PFT, sputum, CT will be done at baseline, 18mo and 36 mo.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris-Gimbel, MD, MS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Montefiore Hospital, CTRC MUH, Keystone Bldg., Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Gingo MR, Nouraie M, Kessinger CJ, Greenblatt RM, Huang L, Kleerup EC, Kingsley L, McMahon DK, Morris A. Decreased Lung Function and All-Cause Mortality in HIV-infected Individuals. Ann Am Thorac Soc. 2018 Feb;15(2):192-199. doi: 10.1513/AnnalsATS.201606-492OC. PMID 29313714